CLINICAL TRIAL: NCT02877667
Title: Soliton Planar Acoustic Wave Device System for Dermal Clearing Human Trial Protocol
Acronym: SOL1601
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soliton (Industry)
Collaborators: MedSource LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soliton 2016-001
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Tattoo
Keywords: tattoo; laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label device treatment (Experimental): Up to four passes with Q-Switched laser alternating with acoustic wave device
  Interventions: Device: planar acoustic wave device

INTERVENTIONS:
Device: planar acoustic wave device — accessory to laser treatment
  Other Names: AWD

SUMMARY:
Study of new acoustic wave device as an accessory to laser treatment in tattoo reduction.

DETAILED DESCRIPTION:
A non-significant risk, single center, prospective device trial to evaluate the number of passes of Q-Switch laser treatment that can be completed with a Q-Switch Laser alone compared to use of the Soliton Planar Acoustic Wave Device System (AWD) System as an accessory to Q-switched laser in tattoo reduction treatment.

ELIGIBILITY:
Inclusion Criteria:

* Range of Fitzpatrick skin color scores I to III
* Tattoo with location on arms, legs, and torso only, and accessible to AWD treatment head. Black ink only. Other ink colors may be present, but areas of black only tattoo should meet criteria described as: minimum 1" x 3" tattoo with at least 30-50% consistent coverage (see fig 1).
* Tattoo age between 1 and 20 years.
* Professionally applied.

Exclusion Criteria:

* Subject is pregnant or planning to become pregnant during the duration of the study.
* Prior tattoo removal procedures on target tattoo.
* Self-applied or amateur tattoo.
* Tattoo layering (additional tattoo placed over an older tattoo to hide it) on target tattoo.
* Metal or plastic implants in the area of the tattoo (pacemaker, implanted defibrillator, stent, or implants in the hips, knees, elbows, etc.).

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Demonstrate that multiple passes with Quality Switched Yag laser is safe based on assessment of Adverse Events | 1 day
  Safety assessments included reported Adverse Events as a result of physician examination

SECONDARY OUTCOMES:
Efficacy comparison of tattoo fading of laser versus laser and Acoustic Wave Device treated tattoos . | 12 weeks
  The degree of fading assessed in terms of percentage fading (1-100%) and according to the following 1 to 5 scale:
  * 1 = 0%;
  * 2 = 1-25%;
  * 3 = 26-49%;
  * 4 = 50-75%; or
  * 5 = 76-100%

CONTACTS AND LOCATIONS:
Overall Officials: Chris Capelli, MD, Study Director — Soliton
Locations (1):
- SkinCare Physicians, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No